CLINICAL TRIAL: NCT05070507
Title: Preventive Effect of an Enzyme-containing Lozenge on Dental Biofilm Accumulation in Healthy Individuals: A Clinical Pilot Study.
Brief Title: Effect of an Enzyme-containing Lozenge on Dental Biofilm in Healthy Individuals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novozymes A/S (Industry)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NZ-OHBFC-2020-04
Record Dates: First submitted 2021-09-12; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Dental Plaque; Gingivitis; Microbial Colonization
MeSH Terms: conditions — Dental Plaque; Gingivitis; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enzyme containing lozenge (Experimental)
  Interventions: Dietary Supplement: Enzyme containing lozenge
- Placebo lozenge (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo lozenge

INTERVENTIONS:
Dietary Supplement: Enzyme containing lozenge — Subjects are instructed to take one lozenge three times daily, at least 30 minutes after a meal, for seven days. No oral health care procedures are allowed during the intervention period.
  Arms: Enzyme containing lozenge
Dietary Supplement: Placebo lozenge — Subjects are instructed to take one lozenge three times daily, at least 30 minutes after a meal, for seven days. No oral health care procedures are allowed during the intervention period.
  Arms: Placebo lozenge

SUMMARY:
The purpose of the study is to assess the effect of an enzyme containing lozenge on dental plaque accumulation in healthy adults.

DETAILED DESCRIPTION:
The purpose of this study is to examine the clinical effects of a lozenge containing enzymes on dental plaque accumulation and oral microbiome composition after professional dental cleaning, as compared to a placebo lozenge without enzymes. Furthermore, safety of the enzyme lozenge will be assessed by clinical evaluation of the oral hard and soft tissues. The null hypothesis is that the treatment with enzyme-containing lozenges do not affect plaque accumulation, as compared to a placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy males and females ≥18 years of age.
* Able to read, sign and receive a copy of the signed informed consent form.
* Have at least 20 natural teeth.

Exclusion Criteria:

* Clinically visible active caries lesions and/or periodontitis.
* Significant oral soft tissue pathology based on a visual examination.
* History of allergy or significant adverse events following use of oral hygiene products such as toothpastes, mouth rinses, breath mints, lozenges, or chewing gum or their ingredients.
* History of allergies to ingredients in the test product.
* History of allergies towards enzymes.
* Self-reported as pregnant or nursing.
* Self-reported serious medical conditions.
* Antibiotic or anti-inflammatory medication within 30 days of screening visit.
* Orthodontic appliances, including retainers, peri/oral piercings, or removable partial dentures.
* Acute sinusitis or severe oral-pharyngeal infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Accumulation of dental plaque after 24 hours | Change in dental plaque score from baseline to 24 hours' follow-up
  Dental plaque assessed by the modified Quigley-Hein Plaque Index

SECONDARY OUTCOMES:
Accumulation of dental plaque after 7 days | Change in dental plaque score from baseline to 7 days' follow-up
  Dental plaque assessed by the modified Quigley-Hein Plaque Index
Development of gingivitis after 7 days | Change in gingivitis score from baseline to 7 days' follow-up
  Gingivitis assessed by the Silness-Löe Plaque Index
Microbial characterization of the oral microbiome from plaque and saliva samples | 7 days' follow-up
  Assessed by 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Schlafer, DDS, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No